CLINICAL TRIAL: NCT03473184
Title: A 4 Day, Randomized Study to Evaluate the Potential of CCP-020 (Diacerein 1%) Topical Ointment to Induce a Phototoxicity Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test
Brief Title: A 4-Day Study to Evaluate the Photoxicity of Diacerein 1% Topical Ointment in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Castle Creek Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCP-020-104
Record Dates: First submitted 2018-03-05; First posted 2018-03-22 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — diacerein; Ointments

STUDY DESIGN:
Intervention Model Description: Phototoxicity Potential Assessment (Photopatch test). All subjects received applications of 0.2 mL of diacerein 1% ointment and vehicle ointment under occlusive patch conditions to 2 skin sites at the infrascapular area of the back for approximately 24 (±2) hours. Following the removal of the patches, one site was irradiated and one remained non-irradiated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Cohort (Healthy Volunteers) (Experimental): Single cohort received diacerein 1% ointment
  Interventions: Drug: Diacerein 1% ointment

INTERVENTIONS:
Drug: Diacerein 1% ointment — Diacerein 1% ointment and vehicle ointment were applied on Day 1 at two randomly assigned skin sites on each side of the lower thoracic area of the back according to a randomization scheme. One side of the back was irradiated on Day 2, including an untreated irradiated control site, and the other side was to remain non-irradiated.
  Other Names: CCP-020

SUMMARY:
This study was designed to assess the phototoxic potential of diacerein 1% ointment when application is followed by light exposure.

DETAILED DESCRIPTION:
This was a single-center, randomized, within-subject comparison of diacerein 1% ointment and vehicle ointment applied to 2 sites on opposite sides of the the infrascapular area of the back under occlusive patch conditions for approximately 24 (±2) hours. Product was applied according to the randomization scheme in an amount of 0.2 mL, once during the study.

Patches were removed and 1 of the skin sites for each product was irradiated and 1 remained non-irradiated. The irradiated and non-irradiated sites were compared with each other and with an untreated irradiated control site.

ELIGIBILITY:
Key Inclusion Criteria:

* Is a healthy male or female (to be confirmed by medical history);
* Is 18 years of age or older;
* In the case of a female of childbearing potential, is using two acceptable forms of birth control;
* In the case of a female of childbearing potential, has a negative urine pregnancy test (UPT) at Day 1 and are willing to submit to a UPT at the end of study (EOS);
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events (AEs);
* Is of any Fitzpatrick Skin Type or race, providing the skin pigmentation will allow discernment of erythema

Key Exclusion Criteria:

* Has a history of photosensitivity or photoallergy;
* Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction;
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study, or systemic/topical antihistamines 72 hours prior to and during the study;
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics such as aspirin (occasional use of acetaminophen will be permitted);
* Is taking medication known to cause phototoxic reactions (eg, tetracyclines, thiazides, nonsteroidal anti-inflammatory drugs [NSAIDs]);
* Has psoriasis and/or active atopic dermatitis/eczema;
* Has known sensitivity or allergy to constituents of materials being evaluated including diacerein, mineral oil, petrolatum, cetyl alcohol, D&C Yellow #10 and/or ethyl paraben;
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans,uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* Has received treatment for any type of internal cancer within 5 years prior to study entry;
* Has any known sensitivity to adhesives; and/or
* Has received any investigational drug(s) within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Spellman, MD, Study Chair — Castle Creek Pharmaceuticals, LLC
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: skin sites
Groups:
- Single Cohort (Healthy Volunteers): Diacerein 1% ointment and vehicle ointment were applied on Day 1 at two randomly assigned skin sites on each side of the lower thoracic area of the back according to a randomization scheme. One side of the back was irradiated on Day 2, including an untreated irradiated control site, and the other side was to remain non-irradiated.
Period: Overall Study
Arm/Group | Single Cohort (Healthy Volunteers)
Started | 34; 170 skin sites
Diacerein 1% Ointment Irradiated | 34; 34 skin sites
Vehicle Ointment Irradiated | 34; 34 skin sites
Diacerein 1% Ointment Non-irradiated | 34; 34 skin sites
Vehicle Ointment Non-irradiated | 34; 34 skin sites
Untreated Irradiated | 34; 34 skin sites
Completed | 34; 170 skin sites
Not Completed | 0; 0 skin sites

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort (Healthy Volunteers)
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 55.0 [23 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Observed Phototoxicity
Description: The mean of the total irritation scores 24 and 48 hours post the site irradiation procedure. ( i.e. Day 3 and 4) Total Irritation Score is a visual score summing the degree of erythema and edema. Minimum score= 0; Maximum score = 5; higher score = worse outcome.
Time Frame: Days 3 and 4 (24 and 48 hours post site irradiation procedure)
Population: 5 skin sites on each of 34 participants for a total of 170 skin sites evaluated.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: skin sites
Groups:
- Single Cohort (Healthy Volunteer): Diacerein 1% ointment and vehicle ointment were applied on Day 1 at two randomly assigned skin sites on each side of the lower thoracic area of the back according to a randomization scheme. One side of the back was irradiated on Day 2, including an untreated irradiated control site, and the other side was to remain non-irradiated.
Arm/Group | Single Cohort (Healthy Volunteer)
Number analyzed (Participants) | 34
Number analyzed (skin sites) | 170
Score on a scale
  Diacerein 1% ointment irradiated: number analyzed (skin sites) | 34
  Diacerein 1% ointment irradiated | 0.15 (0.31)
  Vehicle ointment irradiated: number analyzed (skin sites) | 34
  Vehicle ointment irradiated | 0.15 (0.31)
  Diacerein 1% ointment non-irradiated: number analyzed (skin sites) | 34
  Diacerein 1% ointment non-irradiated | 0.00 (0.00)
  Vehicle ointment non-irradiated: number analyzed (skin sites) | 34
  Vehicle ointment non-irradiated | 0.00 (0.00)
  Untreated irradiated: number analyzed (skin sites) | 34
  Untreated irradiated | 0.15 (0.31)
Statistical Analysis 1: Comparison: Single Cohort (Healthy Volunteer); Irradiated vehicle and untreated irradiated sites versus irradiated diacerein site, and non-irradiated vehicle site versus non-irradiated diacerein site and untreated irradiated site versus irradiated vehicle site; Test type: Other — p-values are from an ANOVA of the average numerical score (sum of erythema and edema) at 24 and 48 hours post irradiation (Days 3 and 4) with effects of subject and treatment, using Fisher's least significant differences; p = 1.0000, ANOVA
Statistical Analysis 2: Comparison: Single Cohort (Healthy Volunteer); Non-irradiated diacerein and vehicle sites versus irradiated diacerein site, and irradiated vehicle and untreated irradiated sites versus non-irradiated diacerein site, and non-irradiated vehicle site versus irradiated vehicle site, and untreated irradiated site versus non-irradiated vehicle site; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0008, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were to be reported from first dose through completion of the last study visit (i.e. Four days).
Description: Adverse events were not assessed at a patch site-specific level.
Arm/Group | Single Cohort (Healthy Volunteers)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT03473184/Prot_SAP_000.pdf